CLINICAL TRIAL: NCT04254458
Title: Laser Peripheral Iridotomy Induced Changes in Corneal Densitometry in Acute Primary Angle Closure Glaucoma Cases
Brief Title: Corneal Densitometry in Acute Primary Angle Closure Glaucoma
Status: Completed | Type: Observational
Sponsor: Ulucanlar Eye Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ufuk Elgin, Professor, Ulucanlar Eye Training and Research Hospital
Other Study IDs: E-18-1866
Record Dates: First submitted 2020-01-29; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Acute Primary Angle-closure Glaucoma
Keywords: Cornea,; density,; laser peripheral iridotomy,; primary angle closure glaucoma
MeSH Terms: conditions — Corneal Diseases; Glaucoma, Angle-Closure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PACG group: Cases who had first acute attack of primary angle closure glaucoma
  Interventions: Diagnostic Test: Corneal densitometry

INTERVENTIONS:
Diagnostic Test: Corneal densitometry — Corneal density values were measured by densitometry software of Pentacam HR-Scheimpflug corneal topography

SUMMARY:
Purpose: Our purpose was to investigate the laser peripheral iridotomy (LPI) induced changes in corneal densitometry in acute primary angle closure glaucoma (PACG) cases during the post-laser 1 month period.

Material and methods: This prospective study included 21 eyes of 21 cases with first acute attack of PACG. All the eyes underwent LPI with neodymium: yttrium-aluminum-garnet (Nd: YAG) laser after the intraocular pressure (IOP) decreased to normal levels with maximal systemic and topical anti-glaucoma treatment and complete regression of clinically significant corneal edema. Central corneal thickness (CCT) and corneal density values were measured by densitometry software of Pentacam HR-Scheimpflug corneal topography over a 12-mm diameter of the cornea just before LPI and at the first week and the first month after LPI. Kolmogorov smirnov and paired-t tests were used for statistical analysis.

DETAILED DESCRIPTION:
This prospective study included 21 eyes of 21 cases with first acute attack of PACG who had applied to emergency department of Ulucanlar Eye Research Hospital between March 2018 and January 2019. All the eyes underwent LPI with neodymium: yttrium-aluminum-garnet (Nd: YAG) laser after the IOP decreased to normal levels with maximal systemic and topical anti-glaucoma treatment and complete regression of clinically significant corneal edema.

During the acute attack ocular examination was performed at the emergency department including best-corrected visual acuity (BCVA) with Snellen charts, slit-lamb examination, fundus examination by +90 D lens, IOP measurements with Goldmann applanation tonometry, gonioscopy of the fellow eye with Goldmann three-mirror lens. Gonioscopy and fundus examinations were performed for the eyes with acute PACG after the regression of corneal edema.

All the cases had intravenous infusion of mannitol 20% (250-300 cc) at the emergency department. Oral acetazolamide 250 mg (3 times daily), oral potassium supplement, topical fixed-combination of beta-blocker and carbonic anhydrase inhibitors (twice daily) and brimonidine (twice daily). LPI procedures were performed within the first day of the attack (after 12-24 hours) by the same experienced physician (OA) with neodymium: yttrium-aluminum-garnet (Nd: YAG) laser under topical anesthesia with proparacain %0.5. Superior-nasal position (1 or 11 o'clock) was focused and 1 or more shots were performed (1-3 pulses per shot with 3-8 mJ energy).

Central corneal thickness (CCT) and CD values were measured by densitometry software of Pentacam HR-Scheimpflug corneal topography just before LPI and at the first week and the first month after LPI. All the measurements were performed by the same experienced clinician between 9 am and 2 pm under standard dim-light conditions without pupil dilatation.

ELIGIBILITY:
Inclusion Criteria:

* Acute primary angle closure glaucoma cases with first attack
* high IOP (>40 mmHg)
* corneal edema
* red eye
* mid-dilated pupil
* presence of the symptoms like blurred vision, halos, ocular pain, headache, nausea and vomiting

Exclusion Criteria:

* The cases who had histories of any types of glaucoma or increased IOP before
* any corneal diseases like keratokonus
* corneal opacity
* dry eye or any ocular surface diseases
* ocular surgery or laser treatment
* trauma
* uveitis or other inflammation and contact lens use and diabetic cases were excluded

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients were Turkish Caucasians with with first attack of primary angle closure glaucoma
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Measurement of corneal density by Pentacam HR-Scheimpflug corneal topography | 1 month
  The measurements were done between 9 am and 2 pm under standard dim-light conditions without pupil dilatation. The CD values of anterior layer (anterior 120 µm), central (between anterior layer and posterior 60 µm), posterior layer (posterior 60 µm) of 4 annular concentric zones as 0-2 mm zone, 2-6 mm zone, 6-10 mm zone and 10-12 mm zone were measured. The CD values were expressed in grayscale units (GSC) as 0 for maximum transparency and 100 for total corneal opacity. Measurement were done just before laser treatment and repeated at the first week and month.

SECONDARY OUTCOMES:
Measurement of central corneal thickness by Pentacam HR-Scheimpflug corneal topography | 1 month
  The measurements were done between 9 am and 2 pm under standard dim-light conditions without pupil dilatation. The central corneal thickness measurements just before laser treatment and at the first week and the first month.

CONTACTS AND LOCATIONS:
Locations (1):
- Ufuk Elgin, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No